CLINICAL TRIAL: NCT01441492
Title: A Randomized Prospective Multicenter Trial of Pancreas Resection With and Without Routine Intraperitoneal Drainage
Brief Title: Pancreas Resection With and Without Drains
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, William E Fisher, Director, Elkins Pancreas Center, Professor, Michael E. DeBakey Department of Surgery, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-28324
Record Dates: First submitted 2011-09-23; First posted 2011-09-27 (Estimated); Results first posted 2020-08-31 (Actual); Last update posted 2020-08-31 (Actual); Status verified 2020-08

CONDITIONS: Pancreas Tumor; Pancreatitis
Keywords: Distal pancreatectomy; Pancreas resection
MeSH Terms: conditions — Pancreatic Neoplasms; Pancreatitis | interventions — Drainage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- No Drains (Experimental): Patients who will not receive intraperitoneal drainage following pancreas resection.
  Interventions: Procedure: No Drains
- Drains (Experimental): Patients who will receive drains, the standard of care treatment, following pancreas resection.
  Interventions: Procedure: Drains

INTERVENTIONS:
Procedure: No Drains — A closed-suction drain will not be placed near the transection margin at the time of surgery in the experimental group.
  Arms: No Drains
Procedure: Drains — A drain will be placed near the pancreatic transection margin at the time of surgery (standard of care).
  Other Names: The specific brand of drain is not contolled.
  Arms: Drains

SUMMARY:
This randomized prospective trial is designed to test the hypothesis that pancreatectomy without routine intraperitoneal drainage does not increase the severity or frequency of complications within 60 days of surgery.

DETAILED DESCRIPTION:
The rate of pancreatic fistula after pancreas resection is about 10% and surgeons have traditionally placed drains near the pancreatic anastomosis to control this potentially very serious complication. In recent years, advances in interventional radiology have allowed safe percutaneous drainage of intra-abdominal fluid collections. Some surgeons have abandoned the routine use of prophylactic drains placed at the time of pancreas resection and rely on percutaneous drainage for the minority of patients who develop a pancreatic fistula.

Hypothesis:

This randomized prospective trial is designed to test the hypothesis that pancreatectomy without routine intraperitoneal drainage does not increase the severity or frequency of complications within 60 days of surgery. The primary endpoint to assess the severity of complications will be the number of patients with any ≥ Grade II complication. Severity of complications experienced will also be assessed by comparing the number of patients with, any ≥ Grade III complication, any serious adverse event (SAE), and the median complication severity grade of all complications. The frequency of complications will be assessed by comparing the number of patients with 1, 2, 3, 4, 5, or more than 5 complications of any severity grade.

Objectives:

Primary: Difference in 60-day ≥ Grade II complication rate comparison between patients who receive a pancreatectomy without routine intraperitoneal drainage and those who do receive routine intraperitoneal drainage.

Secondary:

A. 60-day ≥ Grade III complication rate comparison between patients who receive a pancreatectomy without routine intraperitoneal drainage and those who do receive routine intraperitoneal drainage.

B. Serious adverse event (SAE) rate comparison between patients who receive a pancreatectomy without routine intraperitoneal drainage and those who do receive routine intraperitoneal drainage.

C. Median complication severity grade comparison between patients who receive a pancreatectomy without routine intraperitoneal drainage and those who do receive routine intraperitoneal drainage.

D. 60-day frequency of complications (any Grade) between patients who receive a pancreatectomy without routine intraperitoneal drainage and those who do receive routine intraperitoneal drainage.

E. 60-day, and 90-day mortality rate comparison between patients who receive a pancreatetomy without routine intraperitoneal drainage and those who do receive routine intraperitoneal drainage.

F. Rate of specific complications compared between patients who receive a pancreatectomy without routine intraperitoneal drainage and those who do receive routine intraperitoneal drainage.

G. Length of stay (index admission and total within 60 days) comparison between patients who receive a pancreatectomy without routine intraperitoneal drainage and those who do receive routine intraperitoneal drainage.

H. Crude cost comparison between patients who receive a pancreatectomy without routine intraperitoneal drainage and those who do receive routine intraperitoneal drainage.

I. Quality of life comparison between patients who receive a pancreatectomy without routine intraperitoneal drainage and those who do receive routine intraperitoneal drainage.

ELIGIBILITY:
Inclusion Criteria:

* The subject has a surgical indication for distal pancreatectomy.
* In the opinion of the surgeon, the subject has no medical contraindications to pancreatectomy.
* At least 18 years of age.
* The subject is willing to consent to randomization to the intraperitoneal drain vs. no drain group.
* The subject is willing to comply with 90-day follow-up and answer quality-of-life questionnaires per protocol.

Exclusion Criteria:

* The subject does not have a surgical indication for distal pancreatectomy.
* In the opinion of the surgeon, the subject has medical contraindications to pancreatectomy.
* Less than 18 years of age.
* The subject is not willing to consent to randomization to the intraperitoneal drain vs. no drain group.
* The subject is not willing to comply with 90-day follow-up and answer quality-of-life questionnaires per protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 399 (Actual)
Dates: Start 2011-09; Primary Completion 2016-09 (Actual); Study Completion 2017-07-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William E Fisher, MD, Principal Investigator — Baylor College of Medicine
Locations (14):
- United States (12):
  - University of Florida Health, Gainesville, Florida
  - University of South Florida, Tampa, Florida
  - Indiana University - Purdue University Indianapolis, Indianapolis, Indiana
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Winthrop-University Hospital, Mineola, New York
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Tennessee Health Science Center, Memphis, Tennessee
  - University of Texas Medical Branch, Galveston, Texas
  - Baylor College of Medicine, Houston, Texas
- Canada (2):
  - University of Calgary, Calgary, Alberta
  - Sunnybrook Health Sciences Centre, Toronto, Ontario

REFERENCES:
- [Background] Fisher WE, Hodges SE, Silberfein EJ, Artinyan A, Ahern CH, Jo E, Brunicardi FC. Pancreatic resection without routine intraperitoneal drainage. HPB (Oxford). 2011 Jul;13(7):503-10. doi: 10.1111/j.1477-2574.2011.00331.x. PMID 21689234
- [Background] Van Buren G 2nd, Bloomston M, Hughes SJ, Winter J, Behrman SW, Zyromski NJ, Vollmer C, Velanovich V, Riall T, Muscarella P, Trevino J, Nakeeb A, Schmidt CM, Behrns K, Ellison EC, Barakat O, Perry KA, Drebin J, House M, Abdel-Misih S, Silberfein EJ, Goldin S, Brown K, Mohammed S, Hodges SE, McElhany A, Issazadeh M, Jo E, Mo Q, Fisher WE. A randomized prospective multicenter trial of pancreaticoduodenectomy with and without routine intraperitoneal drainage. Ann Surg. 2014 Apr;259(4):605-12. doi: 10.1097/SLA.0000000000000460. PMID 24374513
- See also: Elkins Pancreas Center — https://www.bcm.edu/healthcare/care-centers/pancreas-center

RESULTS

PARTICIPANT FLOW:
Groups:
- No Drains: Patients did not receive intraperitoneal drainage following pancreas resection.
  No Drains: A closed-suction drain was not be placed near the transection margin at the time of surgery in the experimental group.
- Drains: Patients did receive drain(s), the standard of care treatment, following pancreas resection.
  Drains: A drain was placed near the pancreatic transection margin at the time of surgery (standard of care).
Period: Overall Study
Arm/Group | No Drains | Drains
Started | 197 | 202
Completed | 170 | 174
Not Completed | 27 | 28

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | No Drains | Drains | Total
Number analyzed (Participants) | 170 | 174 | 344
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 60 [47 to 73] | 61 [49 to 73] | 61 [48 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103 | 102 | 205
  Male | 67 | 72 | 139
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 5 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 17 | 25 | 42
  White | 126 | 123 | 249
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 23 | 21 | 44

OUTCOME MEASURES:

1. Primary Outcome: 60-day ≥ Grade II Complication Rate
Description: The primary outcome measure was defined as the number of patients with grade 2 or higher grade complications within 60 days of the date of surgery will be meticulously recorded using specific and standardized definitions. Complications will be graded in severity using the Common Terminology Criteria for Adverse Events CTCAE (v4.0) (Grade 1-5) unless otherwise stated below. For grading schemes with A, B, C rather than 1-5, severity scores will be converted to 1-3.
Time Frame: 60 days
Measure: Count of Participants; unit: Participants
Arm/Group | No Drains | Drains
Number analyzed (Participants) | 170 | 174
Participants | 72 | 76
Statistical Analysis 1: Comparison: No Drains vs Drains; the study is powered to be able to detect a 15% difference in the ≥ Grade II complication rate between the drain and no drain groups. A total of 342 evaluable patients will be needed for the two study groups (n=171 per group) in order to achieve 80% power to detect a 15% increase or decrease in the complication rate with a significance level of 0.05; Test type: Other; p = 0.804, Chi-squared

2. Secondary Outcome: 60-day ≥ Grade III Complication Rate
Description: This secondary outcome measure was defined as the number of patients with one or more complications with grade 3 or higher grade within 60 days of the date of surgery. Complications will be graded in severity suing the Common Terminology Criteria for Adverse Events, CTCAE(v4.0) (Grade 1-5). For grading schemes with A, B, C rather than 1-5, severity scores will be converted to 1-3.
Time Frame: 60 days
Measure: Count of Participants; unit: Participants
Arm/Group | No Drains | Drains
Number analyzed (Participants) | 170 | 174
Participants | 44 | 51

3. Secondary Outcome: Serious Adverse Event (SAE) Rate
Description: This secondary outcome measure is the number of patients with one or more SAE within 60 days of the date of surgery. This outcome will be presented in the Adverse Event Module. The total number of patients affected were 344 (# of no drain=170 vs # of drain=174) and two patients were experienced the serious adverse event (SAE) defined by the protocol. Refer to the Adverse events tables for specifics.
Time Frame: 60 days
Measure: Count of Participants; unit: Participants
Arm/Group | No Drains | Drains
Number analyzed (Participants) | 170 | 174
Participants | 2 | 0

4. Secondary Outcome: Median Complication Severity Grade
Description: This will be calculated for all patients and among just the patients who experienced complications. The complication will be graded in severity using the Common Terminology Criteria for Adverse Events, CTCAE (v4.0) and the severity grade is from 1 to 5. The outcome measure is the median of the Sum of the complication grades of each complication experienced by the patient/# of complications experienced
Time Frame: 60 days
Measure: Median (Inter-Quartile Range); unit: severity grade
Arm/Group | No Drains | Drains
Number analyzed (Participants) | 170 | 174
severity grade
  All patients | 1 [0 to 4] | 1 [0 to 4]
  For just the patients with complications | 4 [2 to 7] | 3 [2 to 6]

5. Secondary Outcome: 60-day Frequency of Complications
Description: This is the median number of complications per patients.
Time Frame: 60 days
Measure: Median (Inter-Quartile Range); unit: Complications per patient
Arm/Group | No Drains | Drains
Number analyzed (Participants) | 170 | 174
Complications per patient | 1 [0 to 2] | 1 [0 to 2]

6. Secondary Outcome: 90-day Mortality Rate
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | No Drains | Drains
Number analyzed (Participants) | 170 | 174
Participants | 2 | 0

7. Secondary Outcome: Rate of Specific Complications
Description: The outcome measure is the number of patients with each particular complication but not including serious adverse events. The complication is using using the Common Terminology Criteria for Adverse Events CTCAE (v4.0).
Time Frame: 60 days
Measure: Count of Participants; unit: Participants
Arm/Group | No Drains | Drains
Number analyzed (Participants) | 170 | 174
Participants
  Pancreatic_leak_fistula | 20 | 88
  Postoperative_Abdominal_FluidCollection | 38 | 15
  Biliary_leak | 1 | 1
  Enteric_leak | 2 | 1
  Lymph_Leak | 1 | 1
  Diarrhea | 17 | 9
  Gastroparesis_DelayedGastricEmptying | 9 | 10
  SmallBowelObstruction | 1 | 3
  Seroma | 3 | 3
  Intra_abd_abscess | 13 | 15
  Wound_Dehiscence | 6 | 4
  Wound_Infection | 5 | 8
  Fever | 36 | 30

8. Secondary Outcome: Length of Stay for the Index Admission
Description: This is the median of length of stay for the index admission. An index admission is an admission in a hospital with a principal diagnosis of a specified condition that meets the inclusion and exclusion criteria for that measure. Total days in the hospital within 60 days of surgery was not collected for analysis. Only length of stay for the index admission was reported.
Time Frame: 60 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | No Drains | Drains
Number analyzed (Participants) | 170 | 174
days | 5 [4 to 6] | 5 [4 to 7]

9. Secondary Outcome: Crude Cost
Description: This is the crude cost of subsequent procedures (CT scan, paracentesis, percutaneous drainage, reoperation) and the length of the index admission and any subsequent readmission. Data were not collected for analysis.
Time Frame: 60 days
Population: Data were not collected for analysis
Arm/Group | No Drains | Drains
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Composite Quality of Life Scores
Description: Subjects will complete the FACT-PA quality of life instrument and the results will be recorded. The quality of life scores at 30 days was collected for analysis.
  The Functional Assessment of Cancer Therapy-Pancreatic Cancer (FACT-PA), is a self-administered pancreas-specific health status survey. The instrument is scored on a scale of 0-28 for Physical well-being subscale(PWB), Social/Family well-being subscale(SWB), Functional well-being subscale(FWB), and on a scale of 0-24 for Emotional well-being subscale(EWB), and on a scale of 0-36 for additional condition of FACT-PA (FACT-PA subscale). The total FACT-G score is the sum of PWB, SWB, FWB, and EWB and the range of 0~108. The total FACT-PA score is the sum of the total FACT-G score and FACT-Pa subscale and the range of 0~144. A lower score represents the worst quality of life.
Time Frame: 30 days and 60 days
Population: The result is the quality of score at 30 days.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | No Drains | Drains
Number analyzed (Participants) | 170 | 174
score on a scale
  Physical well-being subscale | 21 [14 to 27] | 21 [16 to 24]
  Social/Family well-being subscale | 21 [12 to 22] | 21 [18 to 22]
  Emotional well-being subscale | 20 [18 to 23] | 20 [17 to 23]
  Functional well-being subscale | 17 [12 to 22] | 17 [12 to 21]
  Total FACT-G score | 79 [63 to 88] | 79 [66 to 87]
  FACT-Pa subscale | 25 [21 to 28] | 26 [21 to 29]
  Total FACT-Pa score | 104 [84 to 114] | 105 [87 to 116]

ADVERSE EVENTS:
Time Frame: 30 days and 60 days
Arm/Group | No Drains | Drains
Serious Adverse Events (participants affected / at risk) | 2/170 | 0/174
Other Adverse Events (participants affected / at risk) | 99/170 | 130/174
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | No Drains (N=170) | Drains (N=174)
Grade 3 intra-abdominal infection and pancreatic leak/fistula (Surgical and medical procedures) | 2 (2) | 0 (0) — Both SAEs were categorized as grade 3 or higher complications. Both patients were assigned to the "No Drain Group" and developed a grade 3 intra-abdominal infection and pancreatic leak/fistula.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | No Drains (N=170) | Drains (N=174)
Pancreatic_leak_fistula (Gastrointestinal disorders) | 20 | 88
Postoperative_Abdominal_FluidCollection (Gastrointestinal disorders) | 38 | 15
Biliary_leak (Gastrointestinal disorders) | 1 | 1
Enteric_leak (Gastrointestinal disorders) | 2 | 1
Lymph_Leak (Gastrointestinal disorders) | 1 | 1
Diarrhea (Gastrointestinal disorders) | 17 | 9
Gastroparesis_DelayedGastricEmptying (Gastrointestinal disorders) | 9 | 10
SmallBowelObstruction (Gastrointestinal disorders) | 1 | 3
Seroma (Infections and infestations) | 3 | 3
Intra_abd_abscess (Infections and infestations) | 13 | 15
Wound_Dehiscence (Infections and infestations) | 6 | 4
Wound_Infection (Infections and infestations) | 5 | 8
Fever (Infections and infestations) | 36 | 30

LIMITATIONS AND CAVEATS:
A potential weakness of the current study is that it took 5 years to reach targeted accrual.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No